CLINICAL TRIAL: NCT05239611
Title: Feasibility of Home-based Exercise Program for Adults With Cystic Fibrosis to Improve Patient-centered Outcomes, Including a Novel Measure of Ventilation
Brief Title: Feasibility of Home-based Exercise Program for Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00146919
Record Dates: First submitted 2022-01-10; First posted 2022-02-15 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xenon MRI only, without exerercise intervention (Other): Participants will receive usual standard of care and undergo a xenon MRI.
  Interventions: Diagnostic Test: Xenon MRI
- Xenon MRI with exercise coaching (Active Comparator): Participants will receive weekly coaching intervention and undergo a xenon MRI
  Interventions: Diagnostic Test: Xenon MRI

INTERVENTIONS:
Diagnostic Test: Xenon MRI — Study participants will be randomized to a 12 week exercise intervention versus usual care. Participants will have Xenon MRI at study start and completion to evaluate impact of exercise on lung function. The exercise intervention for all participants will be delivered by two pulmonary rehabilitation coaches (PR-coach) including a registered respiratory therapist and clinical registered dietitian who've been trained in exercise training as recommended by the AACVPR and American College of Sports Medicine (ACSM). Each TR participant will be assigned a PR-coach, and receive one weekly exercise consulting session during the 12-week intervention.
  Other Names: exercise

SUMMARY:
The main objective of this clinical pilot study is to evaluate the feasibility and impact of a home-based exercise program on clinical and patient-centered outcomes in adult with cystic fibrosis (CF) and inform the design of a larger clinical trial.

DETAILED DESCRIPTION:
This pilot and feasibility study is a randomized controlled trial comparing exercise intervention with a usual care group. Participants will be randomized based on a randomization table developed by a biostatistician who is not involved in the study. The exercise intervention group will be delivered with a telehealth platform using internet (Zoom HIPAA-Compliant video), an app, phone, and email/text support. Participants will be randomly allocated to either an exercise coaching program or a usual care arm. The exercise intervention arm will follow guidelines established by the American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR) and complement best clinical practices established by the American Thoracic Society/European Respiratory Society (ATS/ERS). The usual care arm will be provided a handout on resources for engaging in physical activity.

Aim 1. Examine the feasibility of a home-based Tele-rehab intervention. Indicators of feasibility will include recruitment and adherence. Hypothesis 1: Based on previous trials, the investigators predict that >50% of eligible participants will consent to the study. Hypothesis 2: Again, based on previous trials, >70% of participants in the intervention arm will adhere to >70% of their weekly prescribed exercise. Also, the investigators will assess reasons for; 1) eligible patients who don't enroll, 2) participants' non-adherence, and 3) non-completers.

Aim 2. Evaluate the impact of a home-based exercise program in adults with CF for improving clinical and patient-centered outcomes. Hypothesis 1: There will be a greater improvement in exercise capacity (measured by a modified shuttle test), a novel measure of lung function 129Xenon MRI (129Xe MRI), forced expiratory volume in 1 second (FEV1), and quality of life with participants in the intervention arm when compared to usual care. Hypothesis 2: Changes in exercise capacity and 129Xe MRI will be associated with exercise adherence, as noted in Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis patients 18 years of age and older, confirmed diagnosis of CF (two CF mutations or sweat chloride > 60 mmol/L)
* stable while either on/off Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) modulator therapy and no plan to start/discontinue CFTR modulator therapy
* clearance from their CF physician to participate in exercise
* have access to the internet
* not involved in an exercise intervention in the previous 6 months, and not performing structured exercise > 150 minutes per week.

Exclusion Criteria:

* pregnancy
* history of solid organ transplant
* active treatment for mycobacterial infections
* significant untreated hypoxemia, oxygen dependent at rest or with exercise
* FEV1 < 40% of predicted or clinical evidence of cor pulmonale
* untreated arterial hypertension (resting systolic blood pressure >140 mm Hg, diastolic blood pressure > 90 mmHg)
* systolic blood pressure less than 90 mm Hg while standing
* congestive heart failure
* active treatment for Allergic Bronchopulmonary Aspergillosis (ABPA)
* acute upper or lower respiratory infection or pulmonary exacerbation within 4 weeks prior to Day 1
* changes in therapy (including antibiotics) for pulmonary disease within 4 weeks prior to Day 1
* significant hemoptysis within 4 weeks prior to Day 1 (≥ 5 mL of blood in one coughing episode or > 30 mL of blood in a 24 hour period
* ongoing participation in an investigational drug study within 60 days prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Burnett, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Pilot participant data available upon request by other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at completion of study analysis. no planned end date
Access Criteria: upon request to primary investigator

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
Started | 9 | 12
Completed | 6 | 8
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Full Range); unit: years] | 28 [24 to 34] | 32 [21 to 49] | 30.6 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 8 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Cardiorespiratory Fitness Assessment- Modified Shuttle Walk Test Result
Description: change in number of modified shuttles completed between baseline/enrollment and study completion at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: change shuttles (1 shuttle is 10 meters)
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
Number analyzed (Participants) | 9 | 12
change shuttles (1 shuttle is 10 meters) | -6.67 (9.33) | -7.63 (9.84)

2. Primary Outcome: Ventilation Defect Percentage (VDP) as Detected by 129Xenon MRI
Description: Hyperpolarized 129Xe ventilation MRI will be performed to assess VDP at baseline (within 2 weeks of initiation of study) and after completion of the intervention/usual care-control period
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of lung with low ventilation
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
Number analyzed (Participants) | 9 | 12
percentage of lung with low ventilation | 20.7 (9.0) | 24.2 (12.6)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second
Description: lung function will be assessed at baseline/enrollment and study completion at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: change pre/post FEV1 percent predicted
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
Number analyzed (Participants) | 6 | 8
change pre/post FEV1 percent predicted | 1.2 (4.66) | -0.38 (3.42)

4. Secondary Outcome: Quality of Life Assessment.
Description: Cystic Fibrosis questionnaire-revised (CFQR) will be assessed at baseline/enrollment and study completion at 3 months. Scale 0-100 (high score indicates better quality of life)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: change pre/post CFQR score
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
Number analyzed (Participants) | 6 | 8
change pre/post CFQR score | -2.0 (10.82) | -4.91 (7.06)

5. Secondary Outcome: Exercise Time
Description: assess weekly adherence to prescribed exercise time completed
Time Frame: 3 months
Population: Participants in the Xenon MRI only without exercise intervention group did not record exercise minutes as they did not have exercise coaching intervention
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Xenon MRI With Exercise Coaching
Number analyzed (Participants) | 12
Minutes | 1290 [285 to 2500]

ADVERSE EVENTS:
Time Frame: study duration, 3 months
Arm/Group | Xenon MRI Only, Without Exerercise Intervention | Xenon MRI With Exercise Coaching
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT05239611/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT05239611/ICF_001.pdf